CLINICAL TRIAL: NCT07399782
Title: EVALUATION OF BOTULINUM TOXIN IN THE PALATOPHARYNGEAL MUSCLE FOR THE TREATMENT OF OBSTRUCTIVE SLEEP APNEA
Brief Title: Botulinum Toxin in the Palatopharyngeal Muscle for the Treatment of Obstructive Sleep Apnea
Acronym: ARAP1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Felicio Rocho (Other)
Responsible Party: Principal Investigator, Alan Rodrigues de Almeida Paiva, Alan Rodrigues de Almeida Paiva, Hospital Felicio Rocho
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90369725.9.0000.5125; 121415 (Other: Hospital Felicio Rocho)
Record Dates: First submitted 2025-08-02; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-08

CONDITIONS: Sleep Apnea Syndrome, Obstructive; Sleep Apnea Syndrome (OSAS); Sleep Apnea/Hypopnea Syndrome; Sleep Apnea - Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Botulinum toxin (Experimental): BOTULINUM TOXIN IN THE PALATOPHARYGEUS MUSCLE
  Interventions: Drug: BOTULINUM TOXIN IN THE PALATOPHARYGEUS MUSCLE

INTERVENTIONS:
Drug: BOTULINUM TOXIN IN THE PALATOPHARYGEUS MUSCLE — Botulinum toxin will be injected into the palatopharyngeal muscle in patients undergoing Medication-Induced Sleep Endoscopy. The injection will be performed while visualizing the posterior pharyngeal constriction.

SUMMARY:
Obstructive Sleep Apnea (OSA) is a sleep-related breathing disorder characterized by recurrent collapse of the upper airway during sleep, in which the palatopharyngeal muscle plays a key role in pathophysiology. Although continuous positive airway pressure (CPAP) remains the standard treatment, adherence is often suboptimal. Botulinum toxin type A (BoNT-A), a peripheral neuromodulator, has been proposed as a potential therapeutic alternative by inducing chemodenervation and muscle volume reduction, thereby potentially increasing upper airway patency. This study aims to evaluate the efficacy and safety of BoNT-A injection into the palatopharyngeal muscle in patients with moderate to severe OSA. This is a prospective, single-arm, interventional clinical trial with pre- and post-intervention assessment. We hypothesize that the intervention will result in a significant reduction in the Apnea-Hypopnea Index (AHI), along with improvements in secondary outcomes such as excessive daytime sleepiness and oxygenation parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe OSA, confirmed by home or laboratory polysomnography.
* Age between 18 and 50 years.
* BMI in the range of 18.5-30.
* Neck circumference ≤ 44 cm (men) and ≤ 42 cm (women).
* Absence of signs of upper obstruction

Exclusion Criteria:

* Skeletal or craniofacial disorders:
* Tonsillar hypertrophy 3-4
* Obesity (BMI > 30 kg/m²)
* Elderly (age > 50 years)
* Neuromuscular diseases (e.g., dystrophies, myasthenia gravis)
* Chronic use of medications that alter muscle tone.
* Excessive alcohol consumption (> 14 drinks/week)
* Chronic obstructive pulmonary disease (COPD)
* Congestive heart failure (NYHA III-IV) or decompensated heart disease.
* Concomitant sleep disorders: narcolepsy, restless legs syndrome, sleep behavior disorder (REM).
* Predominant central or mixed sleep apnea on polysomnography (≥ 50% central events).
* Previous airway surgery (uvulopalatopharyngoplasty, recent tonsillectomy).
* Pregnancy or postpartum (< 6 months).
* Neurological conditions: Previous stroke, Parkinson's disease, dementia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-04-05 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | 12 months
  Evaluate the variation in the Apnea-Hypopnea Index (AHI) before and 3 months after the intervention.

SECONDARY OUTCOMES:
Minimum oxygen saturation (SpO₂) | 12 months
  Verify the impact of the intervention on minimum oxygen saturation (SpO₂)
Epworth Sleepiness Scale | 12 months
  Analyze the change in excessive daytime sleepiness, using the Epworth Sleepiness Scale, before and after the application of botulinum toxin.
Oxygen desaturation index (ODI). | 12 months
  Verify the impact of the intervention on oxygen desaturation index (ODI).

OTHER OUTCOMES:
Adverse events | 12 months
  Monitor the occurrence of adverse events related to the procedure and the application of the toxin, aiming to describe the safety profile of the intervention.

IPD SHARING:
Plan to Share IPD: Yes
Age, Weight, Height, Sex, Test Results, Questionnaire Results, Contact Telephone Number, Intervention Location, Information on Procedures, Procedure Videos
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From the beginning to the end of the study
Access Criteria: Contact the principal investigator via email or phone

REFERENCES:
- [Background] Swislocki ALM, Eisenberg ML. Peyronie Disease as a Marker of Inflammation-Is There Hope on the Horizon? Am J Med. 2021 Oct;134(10):1218-1223. doi: 10.1016/j.amjmed.2021.06.015. Epub 2021 Jul 14. PMID 34273285
- [Result] Dempsey JA, Veasey SC, Morgan BJ, O'Donnell CP. Pathophysiology of sleep apnea. Physiol Rev. 2010 Jan;90(1):47-112. doi: 10.1152/physrev.00043.2008. PMID 20086074